CLINICAL TRIAL: NCT00042783
Title: A Phase II Trial Of A D1/3-MAGE3-HIS Fusion Protein (NSC-719274) With Adjuvant SBAS02B (NSC-719275) For Patients With Stage IV, M1a or M1b Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069468; SWOG-S0116
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: D1/3-MAGE-3-His fusion protein
Biological: SB-AS02B adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Vaccine therapy may be effective in treating stage IV melanoma.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of treating patients with stage IV melanoma with D1/3-MAGE-3-His fusion protein with SB-AS02B adjuvant.
* Determine the clinically confirmed response rates (partial and complete responses) of patients treated with this regimen.
* Determine the 6-month progression-free survival rate of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine immune responses in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive D1/3-MAGE-3-His fusion protein emulsified in SB-AS02B adjuvant intramuscularly once every 3 weeks for a total of 12 weeks (4 injections). In the absence of disease progression or unacceptable toxicity, patients receive a second 12-week course beginning at week 16.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 25-45 patients will be accrued for this study within 5-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma that is considered incurable by surgery, radiotherapy, or limb perfusion

  * M1a or M1b disease
* Measurable disease outside prior field of limb perfusion
* Metastatic mucosal melanoma allowed
* MAGE-3 positive by reverse transcription polymerase chain reaction
* No uveal or choroidal primary melanoma
* No prior or concurrent brain metastases by CT scan or MRI of the brain

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Hepatitis B surface antigen negative
* Hepatitis C negative
* No liver cirrhosis
* No unstable liver disease
* No coagulation disorders

Renal

* Not specified

Cardiovascular

* No major cardiovascular illness
* No myocardial infarction within the past 6 months

Pulmonary

* No major pulmonary illness

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No AIDS or HIV-1-associated complex
* No chronic alcohol abuse or drug addiction
* No systemic infections
* No prior active autoimmune disease
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer from which the patient is currently disease-free

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior adjuvant biologic therapy
* No prior biologic therapy for stage IV melanoma
* No prior MAGE-3 peptide or protein vaccine preparation

Chemotherapy

* At least 4 weeks since prior adjuvant chemotherapy
* No prior chemotherapy for stage IV melanoma

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior adjuvant radiotherapy

Surgery

* At least 4 weeks since prior surgery

Other

* See Disease Characteristics
* At least 3 weeks since prior limb perfusion and recovered
* At least 4 weeks since other prior adjuvant therapy
* No other prior therapy for stage IV melanoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (7):
- United States (7):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - University of Washington School of Medicine, Seattle, Washington